CLINICAL TRIAL: NCT05562128
Title: Effects of Forest Therapy on Physical and Psychological Parameters in the General Population - a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KWT2
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-12

CONDITIONS: General Population (no Specific Condition or Disease)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active forest therapy (Experimental)
  Interventions: Behavioral: Active forest therapy
- Passive forest therapy (Active Comparator)
  Interventions: Behavioral: Passive forest therapy
- Waiting list (No Intervention)

INTERVENTIONS:
Behavioral: Active forest therapy — Participants take part in a two-hour active clinical forest therapy in Berlin-Wannsee on two days (with a break day in between). In this setting, a trained clinical forest therapist teaches exercises on the perception of nature and the connection between nature and health.
  Arms: Active forest therapy
Behavioral: Passive forest therapy — Participants take part in a two-hour passive clinical forest therapy in Berlin-Wannsee over two days (with a break day in between). In this setting, a trained clinical forest therapist will guide participants to various locations in the forest where participants can stay and let nature have its effect on them.
  Arms: Passive forest therapy

SUMMARY:
In recent years, nature and forest therapy has increasingly become the focus of medical research. Recent scientific findings indicate overall positive effects of nature and forest therapy on physical and mental health. In Asia and Australia, it has already been implemented as a public health concept of prevention and health promotion. The aim of the project is to replicate the experience gained in Asia over the last three decades on the physical and psychological effects of nature/forest therapy in the context of the German forest and to investigate it further scientifically.

ELIGIBILITY:
Inclusion Criteria:

- Ability to Consent

Exclusion Criteria:

* Serious acute or chronic illness
* Immobility or limitation of mobility due to orthopedic, neurologic, or other medical causes
* Participation in another study
* Serious mental illness
* Pregnancy and lactation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | Change from baseline POMS score at 3 months

SECONDARY OUTCOMES:
Profile of Mood States (POMS) | Baseline, day 1, day 3, 1 week, 3 months
Perceived Benefits of Nature Questionnaire (PBNQ) | Baseline, 1 week, 3 months
Subjective Vitality Scale state (SVS-G state) | Baseline, day 1, day 3, 1 week, 3 months
Complaint List (B-LR) | Baseline, 1 week, 3 months
Perceive Stress Questionaire (PSQ) | Baseline, day 1, day 3, 1 week, 3 months
Freiburger Fragebogen zur Achtsamkeit (FFA) | Baseline, 1 week, 3 months
Hospital Anxiety and Depression Scale (HADS) | Baseline, 1 week, 3 months
  The scale ranges from 0 to 3. Higher scores correspond to higher levels of anxiety and/or depression.
Perceived Stress Scale (PSS) | Baseline, 1 week, 3 months
  The scale ranges from 0 to 4. Higher scores correspond to higher levels of perceived stress.
Allgemeine Selbstwirksamkeit Kurzskala (ASKU) | Baseline, 1 week, 3 months
  The scale ranges from 1 to 5. Higher scores correspond to better outcomes.
State-Trait Anxiety Inventory (STAI) | Baseline, day 1, day 3, 1 week, 3 months
  The scale ranges from 1 to 8. Higher scores correspond to higher levels of anxiety (after recoding three inverted items).
PROMIS Scale v1.2 - Global Health | Baseline, 1 week, 3 months
  The scale ranges from 1 to 5, where 1 is the lowest level and 5 is the highest level. Higher scores reflect better functioning.

OTHER OUTCOMES:
Heart Rate Variability (HRV) | Baseline, 1 week
  24h measuring by Faros 180
Qualitative interviews | 1 week and 8 weeks after inclusion
  Qualitative assessment will be carried out in qualitative interviews in 20 patients participating in the study. The interviews will be recorded, transcribed and analyzed with qualitative content analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, State of Berlin, Germany